CLINICAL TRIAL: NCT06805188
Title: Efficacy and Safety of Acupuncture in the Treatment of Osteoarthritis of the Knee: Study Protocol for a Randomized Controlled Trial
Brief Title: Clinical Study of Acupuncture Treatment of Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wu zenan (Other)
Collaborators: The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Wu zenan, Principal Investigator, Jiangxi University of Traditional Chinese Medicine
Organization: Jiangxi University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: JZFYLL20250103002
Record Dates: First submitted 2025-01-16; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis of the Knees; Osteoarthritis (OA) of the Knee; Osteoarthritis
Keywords: Randomized controlled trial; Osteoarthritis of the knee; Acupuncture
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outpatient physicians (X.T and X.Z.X) will perform the initial assessment of the patient, independently enter and collect patient information, and randomize assignment. Patients, outcome assessors and data analysts are not aware of the assignment. The treating physician (W.Z.N) will treat the grouped patients. The statistical analysis team will blind the subgroup assignment and the study. Unblinding will take place at the completion of the trial or at the occurrence of a serious adverse event.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The intervention was performed by two licensed acupuncturists with at least 10 years of clinical experience who received two weeks of training in standardized intervention methods prior to the trial. Acupoints location refers to the WHO Standard Acupuncture Point Locations in the Western Pacific Region (WHO Standard)〔41〕.The acupuncture group will receive the following acupoints (Figure 3, Table 2): the affected side of Chize(LU5), Quchi (LI11), Dubi (ST35), Fengshi (GB31), and Xiyangguan (GB33).
  Interventions: Other: Acupuncture
- Control group (Placebo Comparator): The device's sham needling operation mimics real needling through appearance and tactile sensation, making it difficult for patients to distinguish, meeting the requirement of blinding and effectively controlling the patients' cognitive bias towards the type of intervention. Patients in the sham acupuncture group received this sham acupuncture intervention, which was designed to ensure that only the actual biological effects of acupuncture differed between the experimental group and the control group, and to exclude the psychological implication effects caused by the patients' expectation effects or the operation itself, so as to enhance the scientific validity and reliability of the research results.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture — The intervention was performed by two licensed acupuncturists with at least 10 years of clinical experience who received two weeks of training in standardized intervention methods prior to the trial. Acupoints location refers to the WHO Standard Acupuncture Point Locations in the Western Pacific Region (WHO Standard)〔41〕.The acupuncture group will receive the following acupoints (Figure 3, Table 2): the affected side of Chize(LU5), Quchi (LI11), Dubi (ST35), Fengshi (GB31), and Xiyangguan (GB33).
  Needling was performed with 0.30mm x 40mm disposable Huatuo brand sterile acupuncture needles.After the needles were inserted, needle manipulation was performed at all acupuncture points to achieve the sensations of soreness, numbness, distension, and heaviness.Each acupoint was manipulated for about 30 seconds, and the acupuncture treatment was performed for one 30-minute session.
  Arms: Treatment group
Other: Sham acupuncture — The device's sham needling operation mimics real needling through appearance and tactile sensation, making it difficult for patients to distinguish, meeting the requirement of blinding and effectively controlling the patients' cognitive bias towards the type of intervention. Patients in the sham acupuncture group received this sham acupuncture intervention, which was designed to ensure that only the actual biological effects of acupuncture differed between the experimental group and the control group, and to exclude the psychological implication effects caused by the patients' expectation effects or the operation itself, so as to enhance the scientific validity and reliability of the research results.
  Arms: Control group

SUMMARY:
The main question of this study was to evaluate the efficacy and safety of acupuncture in the treatment of knee osteoarthritis (KOA) through a single-blind, randomized controlled trial divided into two groups. Patients in both groups received a total of 24 acupuncture treatments over an 8-week period. The differences in knee NRS score, WOMAC index, walking test, mental health assessment and other indicators between the acupuncture group and the sham acupuncture group before and after treatment were compared to provide high-quality evidence to support the effectiveness of acupuncture in treating KOA.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a common clinical bone and joint disease.There is a lack of effective specific treatment for KOA.Acupuncture is increasingly being studied for the treatment of KOA, but its efficacy and safety are still controversial.This study aims to provide high-quality evidence by evaluating the results of studies on acupuncture for KOA.

A single-blind, randomized controlled trial design was used in this study, in which the generation and preservation of the randomized sequence was done by an independent follow-up researcher through R software. The random allocation method used was block group randomization to ensure a balanced allocation. At the same time, opaque sealed envelopes containing grouping information were prepared to ensure that the grouping process was concealed. The principle of blinding was strictly implemented throughout the study, and the outcome evaluator was blinded until the end of the trial, when participants remained unknown about their grouping information. The study population consisted of 350 patients with KOA who met the inclusion and exclusion criteria. These patients were randomized in a 1:1 ratio into the following 2 groups:(1) Acupuncture Group (AG) (2) False Acupuncture Group (FAG).Patients in both groups received a total of 24 acupuncture treatments over an 8-week period. The sham acupuncture group utilized a Takakura acupuncture simulation device to mimic acupuncture, where the needles would not penetrate the skin, and the duration of needle retention, treatment points, frequency of treatments, duration of treatment, and follow-up period were kept the same as that of the real acupuncture group. The primary outcome index was the Numerical rating scale (NRS), and secondary outcomes included the Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC),40m Fast-Paced Walking Test(40m FPWT), Roland-Morris Disability Questionnaire (RMDQ), Hamilton Depression Rating Scale (HAMD-17), Hamilton Anxiety Rating Scale (HAMA), Insomnia Severity Index (ISI), Pain self-efficacy questionnaire (PSEQ). Any adverse events during treatment will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years old, regardless of gender
* meeting the diagnostic criteria of the American College of Rheumatology (ACR) of KOA
* patients with an NRS score of at least greater than 4 for knee pain, and the pain has lasted for at least 3 months
* diagnosed with osteoarthritis of the knee by magnetic resonance imaging (MRI) or x-ray in the last 3 years
* volunteering to participate in this trial and signing informed consent

Exclusion Criteria:

* Patients with a history of knee surgery
* Patients who had received any physical therapy related to osteoarthritis of the knee, such as corticosteroid injections, acupuncture, or moxibustion, within the past 3 months
* Patients who had a disease that could lead to pain in the knee, such as a fracture, a synovial cyst, or rheumatoid arthritis
* Patients who had a history of knee surgery. or any significant neurological injury
* Prior serious mental illness, organ failure, or malignancy
* Planned knee surgery within the next 3 months
* Pregnancy or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale | For participants who completed baseline enrollment, efficacy observations were made at treatment enrollment, week 4, week 8, week 16, and week 24.
  The NRS is a commonly used pain assessment tool〔42〕, especially for joint pain, such as knee pain. The scale consists of 11 numbers, ranging from 0 to 10, each representing a different level of pain, and the patient chooses the number that best represents his or her current level of pain according to his or her own pain perception.The NRS score is accurate and concise, and was once regarded as the gold standard for pain assessment by the American Pain Society.

SECONDARY OUTCOMES:
WOMAC index | For participants who completed baseline enrollment, efficacy observations were made at treatment enrollment, week 4, week 8, week 16, and week 24.
  According to the 2020 guidelines for the diagnosis and treatment of osteoarthritis of the knee, four types of indexes are recommended to reflect symptoms and signs, quality of life, structural changes in the joints, and long-term regression. Among them, WOMAC is often chosen as the main outcome index of osteoarthritis index based on the study period, which mainly includes five parts: pain, symptoms, ability to perform activities of daily living, motor function, and quality of life, and the scores can be divided into three grades, and the higher WOMAC index indicates the more serious KOA.
40m FPWT | For participants who completed baseline enrollment, efficacy observations were made at treatment enrollment, week 4, week 8, week 16, and week 24.
  The 40m FPWT for the knee is a test that evaluates knee function, lower extremity muscle strength and walking ability〔44〕. The tester uses a stopwatch or timer to accurately record the total time it takes the subject to complete a 40-meter walk. The shorter the time, the better the subject's knee function, lower limb muscle strength and walking ability.
RMDQ | For participants who completed baseline enrollment, efficacy observations were made at treatment enrollment, week 4, week 8, week 16, and week 24.
  The RMDQ is a questionnaire used to assess functional impairment due to low back pain. The scale consists of 24 items with scores ranging from 0-24, with higher scores indicating more significant functional impairme
Depressive condition | For participants who completed baseline enrollment, efficacy observations were made at treatment enrollment, week 4, week 8, week 16, and week 24.
  Clinically significant depressive symptoms were assessed using the HAMD-17.The HAMD-17 consists of 17 entries, with higher scores indicating more severe depression.
Anxious situation | For participants who completed baseline enrollment, efficacy observations were made at treatment enrollment, week 4, week 8, week 16, and week 24.
  The patients' anxiety symptoms were assessed using the HAMA, which consists of 14 entries, with higher scores indicating more severe anxiety.
Insomnia Severity Index | For participants who completed baseline enrollment, efficacy observations were made at treatment enrollment, week 4, week 8, week 16, and week 24.
  The ISI score was used to assess the sleep quality of the patients.The ISI is an assessment of the status of self-perceived insomnia symptoms in the last two weeks.There are seven items with a total score of 0-28.The higher the score, the more severe the insomnia.
Pain self-efficacy questionnaire | For participants who completed baseline enrollment, efficacy observations were made at treatment enrollment, week 4, week 8, week 16, and week 24.
  PSEQ assesses the impact of pain on patients' daily life, which consists of 10 items scored from 0-60, with higher scores indicating greater self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu Z, Hu Z, Xu Z, Xiao T, Huang Q, Zhou X, Zhang H, Fu Y. Efficacy and Safety of Acupuncture at Sensitized Acupoints for Knee Osteoarthritis: Protocol for a Multicenter, Single-Blind Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 24;14:e77336. doi: 10.2196/77336. PMID 40990366

DOCUMENTS (1):
  • Informed Consent Form (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT06805188/ICF_000.pdf